CLINICAL TRIAL: NCT07279883
Title: Length of Hospital Stay and Postoperative Analgesic Requirements After Introduction of a Specific Maxillary Nerve Block in Children Undergoing Cleft Palate Surgery: a Before-and-after Chart Review Study
Brief Title: Length of Hospital Stay and Postoperative Analgesic Requirements After Introduction of a Specific Maxillary Nerve Block in Children Undergoing Cleft Palate Surgery
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jacob Karlsson, Associate Professor, Karolinska University Hospital
Other Study IDs: Dnr 2025-04058-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cleft Palate Children
Keywords: Cleft palate; Suprazygomatic maxillary nerve block; Pediatric anesthesia; Regional anesthesia; Nerve block; opiod consumtion
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-implementation group (2017): Children who received standard systemic analgesia (intravenous and/or oral opioids, acetaminophen, and NSAIDs) without nerve block.
- Post-implementation group (2018): Children who, in addition to standard systemic analgesia, received a suprazygomatic maxillary nerve block (SZMNB) as part of routine perioperative care.

SUMMARY:
Cleft lip and palate (CLP) is one of the most common congenital malformations and requires repeated surgical correction during childhood. Surgical repair is often associated with significant postoperative pain, traditionally managed with morphine, which carries a risk of undesirable side effects. The suprazygomatic maxillary nerve block (SZMNB) has been shown to provide effective analgesia and may reduce the need for opioids.

Routine use of SZMNB was introduced at the pediatric surgery unit at Karolinska University Hospital in late 2017. A before-and-after evaluation project based on retrospective chart review was initiated in 2018 but was not completed due to the COVID-19 pandemic.

The aim of this project is to investigate whether the introduction of SZMNB has reduced postoperative morphine requirements and opioid-related side effects, and whether this has resulted in shorter hospital stays (earlier discharge) after cleft palate repair.

DETAILED DESCRIPTION:
Scientific background and rationale Cleft lip and palate (CLP) is one of the most common congenital malformations and often requires repeated surgical corrections during childhood. These procedures are associated with considerable postoperative pain that may delay recovery and prolong hospital stay. Traditionally, systemic analgesics (opioids, NSAIDs, and acetaminophen given intravenously or orally) have been used, but these are often insufficient or associated with adverse effects.

Peripheral nerve blocks have become an established and effective method to optimize pain control and reduce side effects in many surgical procedures. The suprazygomatic maxillary nerve block (SZMNB) is a well-described technique that can provide efficient analgesia in cleft palate surgery. Previous studies have demonstrated its safety and analgesic benefits.

Objectives and hypothesis The aim of this study is to evaluate the effectiveness and patient benefits of introducing routine SZMNB as an adjunct to standard analgesic therapy in children undergoing cleft palate surgery at Astrid Lindgren Children's Hospital, Karolinska University Hospital.

Hypothesis: SZMNB provides superior postoperative pain control and shorter hospital stay compared with conventional systemic analgesia alone.

Study design and methods This is a retrospective observational study based on chart review of patients aged 3 months-15 years who underwent cleft palate surgery at Astrid Lindgren Children's Hospital during 2017-2018. No intervention will be performed.

Data will be collected from medical records, including demographics (age, sex, weight), surgical procedure, perioperative and postoperative analgesic regimen (type, dose, timing), presence of SZMNB, pain scores when available, and any recorded adverse effects (nausea, sedation, etc.).

Outcome measures Primary outcome: Length of hospital stay, defined as time from arrival in the recovery unit to the time of discharge documentation.

Secondary outcomes: Total postoperative opioid consumption, need for supplemental analgesia, and frequency of opioid-related side effects (e.g., nausea, sedation).

Statistical analysis Pseudonymized data will be analyzed descriptively and comparatively using standard statistical methods. Results will be presented in tables and figures. Manuscript preparation and analysis will be conducted at Karolinska Institutet, and the results will be submitted for publication in a peer-reviewed journal.

Clinical significance Peripheral nerve blocks such as SZMNB may reduce opioid requirements, shorten hospital stay, and improve recovery in children after cleft palate surgery. This project aims to quantify these effects within our institution. Demonstrated benefits could support wider implementation of SZMNB, improve care efficiency, and enhance the quality of postoperative recovery for affected children.

ELIGIBILITY:
criteria for participating in the study

* children aged 3 months to 15 years.
* Underwent cleft palate (LKG) surgery between 2017-2018.
* Available and complete medical records including perioperative notes, anesthesia documentation, and discharge summaries.
* Received either standard systemic analgesia alone (2017) or standard analgesia plus suprazygomatic maxillary nerve block (SZMNB) (2018).

Exclusion Criteria: not fulfilling inclusion cirteria

-

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of children aged 3 months to 15 years who underwent cleft palate (LKG) surgery at Astrid Lindgren Children's Hospital, Karolinska University Hospital, during 2017-2018.
  All patients received general anesthesia with standard perioperative monitoring and multimodal analgesia. In 2018, a suprazygomatic maxillary nerve block (SZMNB) was introduced as a routine adjunct to systemic analgesia. The study includes two cohorts: one before (2017) and one after (2018) the implementation of SZMNB. Data are collected retrospectively from medical records without any additional interventions.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Through out the study completion, an average of approximately 5 days.
  Time (in hours) from arrival at the postoperative recovery unit to the time of documented discharge by nursing staff in the electronic medical record (TakeCare).

SECONDARY OUTCOMES:
Total postoperative opioid consumption | Through out the study completion, an average of approximately 5 days.
  Total amount of morphine (mg/kg) or morphine-equivalent opioids administered intravenously and/or orally during the postoperative hospital stay.
Need for supplemental analgesia | During postoperative hospital stay.
  Proportion of patients requiring additional rescue analgesics beyond the standard regimen (e.g., extra opioid or NSAID doses).
Incidence of opioid-related side effects | Through out the study completion, an average of approximately 5 days.
  Occurrence of opioid-related adverse effects such as nausea, vomiting, or reduced level of consciousness, as documented in medical records.
Pain scores assessed with validated scale FLACC and VAS | From baseline start of study to after 24 hours.
  Postoperative pain score assessed using FLACC and VAS . High number indicates worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Märit Lundblad, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
This study involves retrospective analysis of patient medical records. Due to Swedish and EU data protection regulations (GDPR), individual participant data cannot be shared publicly. Only aggregated, de-identified summary data will be presented in publications.